CLINICAL TRIAL: NCT05213793
Title: Application of a Noninvasive Quantitative Assessment System for Cerebral Perfusion Function in the "Green Channel" of Acute Stroke
Brief Title: Multi-delay Arterial Spin Labeling Application in Acute Ischemic Stroke
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Xuanwu Hospital, Beijing (Other)
Responsible Party: Principal Investigator, qingfengma, MD, Xuanwu Hospital, Beijing
Other Study IDs: qingfeng ma ASL XuanwuH
Record Dates: First submitted 2022-01-15; First posted 2022-01-28 (Actual); Last update posted 2022-01-28 (Actual); Status verified 2022-01

CONDITIONS: Stroke
Keywords: Ischemic Stroke; Magnetic Resonance Imaging; Cerebrovascular Disease
MeSH Terms: conditions — Stroke; Ischemic Stroke; Cerebrovascular Disorders

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- ischemic stroke: The cohort includes patients with acute stroke who underwent CTP, multi-delay ASL, DWI, CTA or TOF-MRA scanning.All patients will be examined within 24 hours of onset. CBF, CBV, MTT and Tmax cerebral blood flow parameter images of CTP will be obtained. CBF, CBV and ATT cerebral blood flow parameter images in multi-delay ASL will be obtained by the quantitative evaluation system. The volume of reversible ischemic tissue will be calculate according to CTP and multi-delay ASL respectively.
  Interventions: Diagnostic Test: multi-delay arterial spin labeling

INTERVENTIONS:
Diagnostic Test: multi-delay arterial spin labeling — Multi-delay arterial spin labeling is a new method to evaluate the degree of the cerebral perfusion. It can obtain three parameters including CBF,CBV and ATT without radiation,which is similar to the traditional technology. Multi-delay ASL can provide more information of the acute stroke patients.

SUMMARY:
This study explores the value of the non-invasive quantitative evaluation system for cerebral blood flow perfusion function in the diagnosis of stroke. Compared with traditional perfusion techniques, multi-delay arterial spin labeling (ASL) is validated to determine the accuracy of perfusion level, ischemic penumbra and other indexes in patients with acute ischemic stroke. The relationship between perfusion levels of mD-ASL parameters and clinical outcome is also studied.

DETAILED DESCRIPTION:
A total of 200 patients with acute anterior circulation ischemic stroke will be prospectively enrolled.

All patients underwent CTP, multi-delay ASL, DWI, CTA or TOF-MRA scanning. CBF, CBV, MTT and Tmax will be obtained based on CTP, and the range of reversible cerebral ischemia injury will be calculated based on DWI and CTP data. CBF, CBV and ATT images will be obtained based on the multi-delay ASL, and the calculated results of reversible cerebral ischemia injury will also be obtained.

Meanwhile, the image quality of CTP and multi-delay ASL will be evaluated. The time from the patient to the completion of imaging examination and the imaging examination time will be recorded.

Mann-whitney U test and T test can be used to compare the difference of assessment time between different test methods. Chi-square test can be used to compare the differences of image quality among different examination methods. Wilcoxon rank sum test can be used to evaluate the difference between CTP and Multi-delay ASL in terms of parameters and volume of reversible ischemic injury.

ELIGIBILITY:
Inclusion Criteria:

1. Ischemic stroke within 24h；
2. Anterior circulation occlusion confirmed by conventional angiography or magnetic resonance angiography；

Exclusion Criteria:

1. Pregnancy and other contraindication to MRI scan；
2. Informed consent not obtained.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with acute anterior circulation ischemic stroke without contraindication to MRI will be enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2021-04-01 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Compare the volume of reversible ischemic injury of brain tissue measured by multi-delay ASL versus CTP | 24 hours
  Our primary aim is to determine if the diagnostic accuracy of multi-delay Arterial Spin Labeling (ASL) is as good as the diagnostic accuracy of CTP in acute ischemic stroke patient. To test if ASL in noninferior to CTP,

SECONDARY OUTCOMES:
The difference of the procedure of CTP and multi-delay ASL | 24hours
  The researchers will collect the time from diagnosis to completion of imaging examination and the time of imaging examination.Then analyze the time and quality of the multi-delay ASL compared with CTP.

CONTACTS AND LOCATIONS:
Overall Officials: qingfeng Ma, MD, Study Chair — Xuanwu Hospital, Beijing
Locations (1):
- Xuanwu Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Bivard A, Krishnamurthy V, Stanwell P, Levi C, Spratt NJ, Davis S, Parsons M. Arterial spin labeling versus bolus-tracking perfusion in hyperacute stroke. Stroke. 2014 Jan;45(1):127-33. doi: 10.1161/STROKEAHA.113.003218. Epub 2013 Dec 3. PMID 24302482
- [Background] Wang DJ, Alger JR, Qiao JX, Gunther M, Pope WB, Saver JL, Salamon N, Liebeskind DS; UCLA Stroke Investigators. Multi-delay multi-parametric arterial spin-labeled perfusion MRI in acute ischemic stroke - Comparison with dynamic susceptibility contrast enhanced perfusion imaging. Neuroimage Clin. 2013 Jul 6;3:1-7. doi: 10.1016/j.nicl.2013.06.017. eCollection 2013. PMID 24159561